CLINICAL TRIAL: NCT01702207
Title: A One-Year, Prospective, Randomized, Controlled Study Evaluating The Efficacy Of Switching From The Twice Daily Tacrolimus Formulation To The Extended Release, Once Daily Formulation To Reduce The Framingham Cardiovascular Risk Scores.
Brief Title: Evaluation Of Switching From Twice Daily Tacrolimus To Once Daily Formulation On Cardiovascular Risk
Acronym: ESTTEROD
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Saskatchewan (Other)
Collaborators: Astellas Pharma Canada, Inc. (Industry)
Responsible Party: Principal Investigator, AShoker, M.D., University of Saskatchewan
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Supportive Care
Other Study IDs: ESTTEROD
Record Dates: First submitted 2012-09-27; First posted 2012-10-05 (Estimated); Last update posted 2018-01-08 (Actual); Status verified 2018-01

CONDITIONS: Immunosuppression; Cardiovascular Diseases; Kidney Transplantation
Keywords: Prograf®; Advagraf®; tacrolimus; kidney transplant; renal transplant; cardiovascular risk; Framingham Risk; Reynolds Risk; immunosuppression
MeSH Terms: conditions — Cardiovascular Diseases | interventions — Tacrolimus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Once Daily Tacrolimus (Active Comparator): Treatment Arm - Subjects are switched from the tacrolimus twice daily (Prograf®) to the once daily formulation (Advagraf®) to maintain a trough tacrolimus level of 5-8.
  Interventions: Drug: Once Daily Tacrolimus
- Twice Daily Tacrolimus (Active Comparator): Control Arm - Subjects are kept on Prograf® which is the Twice Daily Tacrolimus
  Interventions: Drug: Twice Daily Tacrolimus

INTERVENTIONS:
Drug: Once Daily Tacrolimus — Subjects switched from the tacrolimus twice daily (Prograf®) to the once daily formulation (Advagraf®) to maintain a trough tacrolimus level of 5-8.
  Other Names: Advagraf®
  Arms: Once Daily Tacrolimus
Drug: Twice Daily Tacrolimus — Subjects are kept on Prograf® which is the Twice Daily Tacrolimus
  Other Names: Prograf®
  Arms: Twice Daily Tacrolimus

SUMMARY:
Current standard prophylactic immunosuppression in renal transplantation includes tacrolimus, a calcineurin inhibitor, dosed twice daily. In Canada, oral tacrolimus has been available as a twice daily formulation marketed as Prograf® since 1997. It has recently become available in an extended release formulation called Advagraf®, which is dosed once daily. Advagraf® has been demonstrated to be therapeutically equivalent to Prograf® in the renal transplant maintenance population, and as a result it has been is approved as an alternative to the twice daily formulation in these patients. There is an evolving and expanding positive clinical experience with Advagraf® in kidney transplantation and it has shown to be preferred by many patients, due to the diminished dosing frequency. In clinical trials, Advagraf® has been shown to have other potential benefits over Prograf® such as less inter and intra-patient variability, improved cardiovascular profiles, and improved kidney function. Compared to Prograf®, Advagraf® also has a lower Cmin or 'trough' concentration as well as a lower Cmax or 'peak' concentration. The purpose of this study is to convert stabilized renal transplant patients currently receiving Prograf® to Advagraf®, to investigate these potential therapeutic benefits.

The Framingham Risk Score and the Reynold's Risk Score are currently recommended by the Canadian Cardiovascular Society (CCS) to predict 10-year cardiovascular risk in the general population. Surrogate markers are widely used in clinical trials to shorten follow-up durations. In this study, the investigators will use the Framingham Risk Score and Reynold's Risk Score to quantify changes in estimated cardiovascular risk. The investigators also intend to examine novel inflammatory markers to investigate cardiovascular risk.

The investigators hypothesize that the more consistent drug exposure and lower Cmax noted with Advagraf® will decrease Framingham Risk Score, Reynolds Risk score as well as markers of inflammation in kidney transplant recipients.

ELIGIBILITY:
Inclusion Criteria:

* Kidney transplant patients currently stable on the twice-daily formulation and who are followed as outpatients.
* Stability is defined as change in serum creatinine of less than 10% over the last two months
* Age 18-74 years old
* At least six months after transplantation
* Lack of rejection within the last 12 weeks
* Serum creatinine less than 300 umol/L at enrolment
* Negative urine pregnancy test for female patients of childbearing potential
* Consent to the study
* Not included in a clinical trial within the last 90 days

Exclusion Criteria:

* Patients with other types of solid organ transplants
* Patients with any form of substance abuse or psychiatric disorder.
* Patients with acute or chronic diarrhea
* Patients receiving anti-lymphocyte treatment for rejection within the last six months
* Patients on cyclosporine and or not receiving a mycophenolate derivative.
* Patients with significant liver disease defined as having an elevated bilirubin by at least two times the upper value of the normal range
* Patients who have any unstable medical condition that could interfere with the study
* Patients with chronic viral infection with HIV, Hep C and HCV.
* Presence of any acute illness requiring admission to the hospital for the last 4 weeks
* Pregnancy
* Significant cardiovascular event such as MI, stroke or TIA within the last 12 weeks or uncontrolled hypertension.
* Immunosuppressant changes within the last month.

Ages: 18 Years to 74 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2012-10 (Actual); Primary Completion 2017-12 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
Change in the Framingham risk scores and change in the Reynolds Risk Score. | Visit 1, Visit 3 (12 months)

SECONDARY OUTCOMES:
Comparison in GFR between the two groups. | Visit 1, Visit 3 (12 months)
Effect of therapy on CV biomarkers, insulin resistance and lipid profile. | Visit 1, Visit 3 (12 months)
  CV biomarkers will be assessed by luminex and insulin resistance and lipid profile will be assessed by the Metabolic Syndrome
To look at change in the glomerular filtration rate (GFR) over the duration of the study. | Vist 1, Visit 3 (12 months)

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed Shoker, MD, Principal Investigator — University of Saskatchewan
Locations (1):
- St Paul's Hospital, Saskatoon, Saskatchewan, Canada